CLINICAL TRIAL: NCT03449355
Title: Effect of the Mode of Delivery on Sexual Functions and Quality of Life Among a Group of Egyptian Women
Brief Title: Sexuality After Different Mode of Deliveris
Status: Completed | Type: Observational
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Hanan Nabil, Assistant professor, Mansoura University
Other Study IDs: sexuality
Record Dates: First submitted 2018-02-22; First posted 2018-02-28 (Actual); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: Sexual Dysfunction and the Mode of Deliveries
Keywords: sexuality; mode of delivery; quality of life
MeSH Terms: conditions — Sexual Dysfunction, Physiological; Sexuality

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- vaginal group
- cesarean section group

SUMMARY:
Pregnancy and delivery usually affect the general women's quality of life. Some studies have reported that sexual health may be affected by the mode of delivery. More than 70% of pregnant women prefer C-section due to several reasons point out the fear of pain and complications of vaginal delivery as the most common reasons.

Aim of the work: To explore the relationship between quality of life and the possible sexual dysfunction after normal vaginal in comparison to cesarean section deliveries.

ELIGIBILITY:
Inclusion Criteria:

* Primiparas women who had been delivered by either vaginal or cesarean section about 6-12months.
* All included women should be officially married

Exclusion Criteria:

* Women with history of sexual dysfunction
* Women with history of any pelvic surgery apart from Cesarean.
* history of anti-depressive drug therapy.
* history of genital prolapse
* history of Diabetes mellitus
* loss of any family member or unfaveorouble neonatal outcome or childdeath
* Divorce experience
* family problems and cases who were not interested in participation

Ages: 20 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: primiparous women 6-12 months after deliveries either vaginal or cesarean section
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-01-11 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
quality of life after delivery | one month
  the amplitude of many changes occur during and after pregnancy, which affect physical, psychological and social health and generally women's quality of life

SECONDARY OUTCOMES:
the relationship between quality of life and sexual dysfunction after both modes delivery | one month

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Egypt